CLINICAL TRIAL: NCT05887999
Title: A Phase 1, Randomized, Placebo-Controlled, 2-Period, Cross-over, Double- Blind, Single-Dose Study to Evaluate the Effects of LY3532226 on Insulin- Induced Hypoglycemia in Participants With Type 1 Diabetes Mellitus
Brief Title: A Study of LY3532226 in Participants With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 18064; J2V-MC-GZLC (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-05-25; First posted 2023-06-05 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3532226 (Experimental)
  Interventions: Drug: LY3532226
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3532226 — Administered subcutaneously (SC).
  Arms: LY3532226
Drug: Placebo — Administered SC.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the response of glucagon to insulin-induced low blood sugar after administration of the study drug LY3532226 in participants with type 1 diabetes mellitus (T1DM). The study will also evaluate if LY3532226 helped participants to recover from insulin-induced low blood sugar condition compared to placebo. The study will last approximately 16 weeks excluding screening period.

ELIGIBILITY:
Inclusion Criteria:

* Participants with type 1 diabetes mellitus (T1DM) for at least 2 years treated with insulin
* Body mass index (BMI) of 18.5 to 40.0 kilograms per meter squared (kg/m²)
* Are males or females not of childbearing potential

Exclusion Criteria:

* Have acute proliferative retinopathy requiring active treatment within 3 months of screening
* Have been treated with dipeptidyl peptidase-Ni, GLP-1 receptor agonists, GIP agonists, metformin or sodium-glucose cotransporter 2 inhibitors within the previous 3 months
* Have received systemic or inhaled glucocorticoid therapy
* Women of childbearing potential
* Are currently taking part in another clinical study trial involving medical research, or have participated within the last 30 days of screening in a clinical study involving a study intervention

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamics (PD): Area under the concentration versus time curve from time 60 to 120 minutes (AUC60-120min) of plasma glucagon during the insulin-induced hypoglycemia | Predose up to 120 mins postdose
  PD: AUC60-120min of plasma glucagon during the insulin-induced hypoglycemia

SECONDARY OUTCOMES:
The amount of exogenous glucose infused to maintain a plasma glucose level of >2.5 millimole per liter (mmol/L), after the insulin infusion is terminated. | Predose up to 120 mins postdose
  The amount of exogenous glucose infused to maintain a plasma glucose level of >2.5 mmol/L, after the insulin infusion is terminated.
Change from Baseline in Fasting and Post meal Glucose during Standardized Mixed-meal Tolerance Test (sMMTT) | Predose up to 120 mins postdose
  Change from Baseline in Fasting and Post meal Glucose during sMMTT
Change from Baseline in Glucagon Concentration at Fasting and Post meal during sMMTT | Predose up to 120 mins postdose
  Change from Baseline in Glucagon Concentration at Fasting and Post meal during sMMTT

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- ProSciento, Inc, Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY3532226 in Participants With Type 1 Diabetes Mellitus — https://trials.lilly.com/en-US/trial/407539